CLINICAL TRIAL: NCT03694314
Title: Pilot Study on the Effects of Omega-3 Fatty Acid Supplements on Sleep and Behavior of Mother-child Pairs
Brief Title: Effect of Omega-3 Fatty Acids on Sleep and Behavior (Pilot Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Jianghong Liu, Associate Professor, University of Pennsylvania
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: 829722
Record Dates: First submitted 2018-07-30; First posted 2018-10-03 (Actual); Last update posted 2019-10-08 (Actual); Status verified 2019-10

CONDITIONS: Disturbances in Initiating and Maintaining Sleep; Behavior Problem
Keywords: Omega-3 fatty acids; Sleep; Behavior; Parenting
MeSH Terms: conditions — Mental Disorders; Behavior | interventions — Fatty Acids, Omega-3

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Omega-3 fatty acids (Experimental): Both the mother and child will receive omega-3 supplements in the form of a 200 mL drink to be taken once daily. The intervention will last 45 days. Assessments will take place at 0 months (baseline), 45 days (end of treatment), and 3 months (1 and a half months post-treatment).
  Interventions: Dietary Supplement: Omega-3 fatty acids
- Placebo (Placebo Comparator): The mother and child will both receive a placebo drink to take daily, with no known effect on the brain. The intervention will last 45 days. Assessments will take place at 0 months (baseline), 45 days (end of treatment), and 3 months (1 and a half months post-treatment).
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Omega-3 fatty acids — 200 ml drink. The drink contains 840 mg total of omega-3 (360 mg of DHA, 240 mg of EPA, 200 mg of alpha-linolenic acid, and 40 mg of DPA).
  Arms: Omega-3 fatty acids
Dietary Supplement: Placebo — 200 mL placebo fruit juice with no effect on the hypothesized outcome.
  Arms: Placebo

SUMMARY:
The aim of this feasibility study is to determine whether a nutritional intervention in children and their parents can improve their sleep quality and behavior. The study is a randomized, double-blind, placebo-controlled parallel trial of omega-3 supplementation to children and their mothers.

DETAILED DESCRIPTION:
Previous studies show omega-3 fatty acid supplements improve adolescent's antisocial behavior. However it is less known whether the same effect could be achieved in younger children. Furthermore it is not known whether omega-3 fatty acids could also improve parental behavior and parenting style which could further reduce behavioral problems in children. Moreover, we recently found that children who consume fish more frequently have less sleep problems but it is not known whether omega-3 supplements could also potentially improve children's sleep. We aim to test several hypotheses in this random controlled trial of omega-3 fatty acids.

The study design will consist of a double-blind, randomized placebo-controlled trial of children and their caregivers in a community sample in the city of Philadelphia. It will utilize a random parallel design, in which child and mother pairs will be randomly assigned to either omega-3 supplementation (treatment condition) or a placebo (control condition). This results in 2 groups: (1) child and caregiver both receiving omega-3 and (2) both parent and child receiving the placebo. Treatment will last 45 days. Assessments will take place at 0 months (baseline), 45 days (end of supplementation) and 90 days (45 days after the end of treatment).

ELIGIBILITY:
Inclusion Criteria:

* child between ages 5-9 with mother available to participate in intervention study

Exclusion Criteria:

* intellectual disability
* significant psychiatric and physical illness
* extensive use of nutritional supplements within the past three months
* seafood allergy
* diabetes

Ages: 5 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 29 (Actual)
Dates: Start 2018-05-15 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Sleep | 3 months
  For parent sleep patterns, we will use the Pittsburgh Sleep Quality Index to evaluate changes. For children's sleep, we will use the Child Sleep Habits questionnaire.

SECONDARY OUTCOMES:
Child behavior | 3 months
  Will use the Child Behavior Checklist to evaluate changes in child behavior.
Parental behavior | 3 months
  Will use the Adult Self Report to evaluate changes in parent behavior.
Child and parental cognitive behavior | 3 months
  Will use online cognitive test to evaluate changes in cognition.
Parental style | 3 months
  Will use the Alabama Parenting questionnaire to evaluate changes in parenting style.

CONTACTS AND LOCATIONS:
Overall Officials: Jianghong Liu, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Raine A, Portnoy J, Liu J, Mahoomed T, Hibbeln JR. Reduction in behavior problems with omega-3 supplementation in children aged 8-16 years: a randomized, double-blind, placebo-controlled, stratified, parallel-group trial. J Child Psychol Psychiatry. 2015 May;56(5):509-20. doi: 10.1111/jcpp.12314. Epub 2014 Aug 22. PMID 25146492
- [Background] Liu J, Cui Y, Li L, Wu L, Hanlon A, Pinto-Martin J, Raine A, Hibbeln JR. The mediating role of sleep in the fish consumption - cognitive functioning relationship: a cohort study. Sci Rep. 2017 Dec 21;7(1):17961. doi: 10.1038/s41598-017-17520-w. PMID 29269884